CLINICAL TRIAL: NCT05801068
Title: Effectiveness and Safety of PERIoperative Factor Xa Inhibitor Discontinuation in Patients with Atrial Fibrillation Who Undergoing Minor Bleeding Risk Elective Procedure or Surgery: a Prospective, Multicenter, Noninterventional Study (PERIXa Study)
Brief Title: Perioperative Management of Factor Xa Inhibitors
Acronym: PERIXa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Eue-Keun Choi, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PERIXa
Record Dates: First submitted 2023-03-03; First posted 2023-04-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation; Anticoagulant-induced Bleeding
Keywords: Atrial fibrillation; Perioperative management; Factor Xa inhibitor
MeSH Terms: conditions — Atrial Fibrillation | interventions — Factor Xa Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Periprocedural management of FXa-inhibitor group (Experimental): Hold and resume factor Xa inhibitor during perioperative/periprocedural period according to predefined protocol.
  Interventions: Drug: Factor Xa Inhibitor

INTERVENTIONS:
Drug: Factor Xa Inhibitor — Hold and resume factor Xa inhibitor during perioperative/periprocedural period according to the predefined protocol.
  Other Names: PERIXA group

SUMMARY:
This study aims to analyze the safety and effectiveness of the discontinuation/resumption protocol of factor Xa inhibitors before and after invasive procedures/surgeries in non-valvular atrial fibrillation patients who are at risk of minor bleeding in actual clinical settings

DETAILED DESCRIPTION:
* Study design This is a multicenter, non-randomized, investigator-initiated prospective cohort study. The study will analyze the bleeding risk and incidence of cardiovascular events according to the discontinuation/resumption of factor Xa inhibitors before and after invasive procedures/surgeries in non-valvular atrial fibrillation patients who are prescribed factor Xa inhibitors for stroke prevention and have minor bleeding risk.
* Study population Patients who are over 20 years old, have non-valvular atrial fibrillation, and are taking rivaroxaban, apixaban, or edoxaban (active ingredients), and are facing a procedure defined as having minor bleeding risk.
* Study protocol For patients with non-valvular atrial fibrillation who are prescribed rivaroxaban, apixaban, or edoxaban for stroke prevention and are at risk of minor bleeding, when they visit the prescribing physician (physician A) for consultation and to obtain a medical opinion regarding the discontinuation/resumption of the medication in relation to an invasive procedure, the physician will explain the protocol for discontinuing/resuming the medication and provide a written explanation to ensure that the patient fully understands it.

In addition, the physician in charge of the procedure (physician B) will be notified that the patient has enrolled in this study and will collect information on 1) the type of surgery or procedure performed, and 2) physician B's opinion on the severity of procedure-related bleeding. Thromboembolic and bleeding events will be assessed through patient follow-up 30 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Aged >20 years
* With rivaroxaban, apixaban, or edoxaban
* History of non-valvular atrial fibrillation
* Scheduled minor bleeding risk procedure(s) (dental procedure, cataract/glaucoma surgery, diagnostic GI endoscopy)

Exclusion Criteria:

* Pregnancy
* With rivaroxaban or edoxaban at afternoon
* Mental disorder
* Contraindication to rivaroxaban, apixaban, edoxaban
* Moderate or severe valvular heart disease, or with prosthetic heart valves
* With antiplatelet drugs
* History of systemic embolism or ischemic stroke within the last 12 months
* scheduled therapeutic endoscopic procedure(s)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day major bleeding | Within 30 days after the operation/procedure
  30-day major bleeding

SECONDARY OUTCOMES:
30-day stroke or systemic embolism | Within 30 days after the operation/procedure
  30-day stroke or systemic embolism
30-day death from any cause, stroke or systemic embolism | Within 30 days after the operation/procedure
  30-day death from any cause, stroke or systemic embolism
30-day composite of major bleeding and clinically relevant non major bleeding (CRNMB), and any bleeding | Within 30 days after the operation/procedure
  30-day composite of major bleeding and clinically relevant non major bleeding (CRNMB), and any bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Eue-Keun Choi, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National university Hostpital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwon S, Lee SR, Choi EK, Lee KY, Choi J, Ahn HJ, Oh S, Lip GYH. Perioperative Management in Patients with Atrial Fibrillation Treated with Non-Vitamin K Antagonist Oral Anticoagulants Undergoing Minor Bleeding Risk Procedure: Rationale and Protocol for the PERIXa Study. Vasc Health Risk Manag. 2024 May 17;20:231-244. doi: 10.2147/VHRM.S455530. eCollection 2024. PMID 38774425